CLINICAL TRIAL: NCT00182923
Title: Determinants of Forearm Vascular Relaxation: Role of Genetic Polymorphisms
Brief Title: Forearm Vascular Relaxation
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Other Study IDs: AG0038
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2008-08-29 (Estimated); Status verified 2008-08

CONDITIONS: Healthy
Keywords: Blood pressure; genetics

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to learn the effect of inherited differences on forearm blood flow responses to hormones and drugs

DETAILED DESCRIPTION:
Differences in at least 4 genes are believed to have an important effect on responses to hormones and drugs. For this study, healthy volunteers of normal body weight will be screened to find xxx individuals with the genes of interest. Very small doses of hormones and drugs will be given so that changes in forearm blood flow can be measured, while not causing effects throughout the body. A brachial artery line and venous line will be placed in the study arm so that blood samples may be withdrawn to compare amounts given into the artery and coming out of the vein after circulating through the arm. Forearm blood flow is determined by the rate of swelling of the arm after a blood pressure cuff is inflated (above venous and below arterial blood pressure). The hormones and drugs being studied include angiotensin I, angiotensin II, acetylcholine, sodium nitroprusside, enalaprilat, L-arginine, phenylephrine, endothelin-1, verapamil, and isoproterenol. This procedure will last 4-6 hours. The process will be repeated with the same participant over 2 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Normal physical status without any medical interventions or agents which would alter the defined status of normal

Exclusion Criteria:

* Age less than 21 or greater than 45
* Unable to give informed consent
* BMI (Body Mass Index) less than 18 or greater than 25
* Clinically significant abnormal laboratory values
* Abnormal physical exam
* Abnormal EKG
* Pregnancy
* Smoking or drug usage (illicit or otherwise)
* Post-menopause
* Participation in another clinical trial in the past month
* Chronic Illness

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400
Dates: Start 2003-05; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darrell R. Abernethy, MD, PhD, Principal Investigator — National Institute on Aging, Laboratory of Clinical Investigation
Locations (1):
- National Institute on Aging (NIA), Harbor Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Abernethy DR, Laurie N, Andrawis NS. Local angiotensin-converting enzyme inhibition blunts endothelin-1-induced increase in forearm vascular resistance. Clin Pharmacol Ther. 1995 Sep;58(3):328-34. doi: 10.1016/0009-9236(95)90250-3. PMID 7554707
- [Background] Abernethy DR, Winterbottom LM. Forearm vascular alpha 1-adrenergic blockade by verapamil. Clin Pharmacol Ther. 1990 Jun;47(6):755-9. doi: 10.1038/clpt.1990.104. PMID 2162750
- [Background] Andrawis NS, Craft N, Abernethy DR. Calcium antagonists block angiotensin II-mediated vasoconstriction in humans: comparison with their effect on phenylephrine-induced vasoconstriction. J Pharmacol Exp Ther. 1992 Jun;261(3):879-84. PMID 1602392